CLINICAL TRIAL: NCT00095797
Title: A Phase I Study of XK469R (NSC 698215) in Patients With Refractory Hematologic Malignancies
Brief Title: XK469R in Treating Patients With Refractory Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02633; MDA-2004-0154; U10CA62461 (Other Grant/Funding Number: US NIH Grant/Contract Award Number); CDR0000393836 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Refractory Chronic Lymphocytic Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — XK 469

ARMS (1):
- Treatment (XK469R) (Experimental): Patients receive XK469R IV over 30-60 minutes on days 1, 3, and 5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: R(+)XK469; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: R(+)XK469 — Given IV
  Other Names: XK469
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
Phase I trial to study the effectiveness of XK469R in treating patients who have refractory hematologic cancer. Drugs used in chemotherapy, such XK469R, work in different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicity, maximum tolerated dose, and recommended phase II dose of XK469R in patients with refractory hematologic malignancies.

II. Determine the pharmacokinetics of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the presence of genetic variations potentially affecting XK469R disposition in patients treated with this drug.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive XK469R IV over 30-60 minutes on days 1, 3, and 5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of XK469R until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 6 patients experience dose-limiting toxicity. A total of 12 patients receive treatment at the MTD.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following relapsed or refractory hematologic malignancies for which all potentially curative therapy options have been exhausted:

  * Acute myeloid leukemia* (AML) (non-M3)
  * Acute lymphoblastic leukemia*
  * Myelodysplastic syndromes*, including the following:

    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
  * Chronic myelomonocytic leukemia in transformation* (CMML-t) with ≥ 10% peripheral blood/bone marrow blasts
  * Chronic myelogenous leukemia in blast crisis* (CML-BC)
  * Chronic lymphocytic leukemia

    * Rai stage III-IV
    * Failed prior fludarabine-based therapy and ≥ 1 other therapy

      * Fludarabine failure defined as failure to achieve partial response or complete response (CR) to at least 1 fludarabine-containing regimen; disease progression while on fludarabine; or disease progression within 6 months of response to fludarabine
* Not a candidate for autologous or allogeneic stem cell transplantation (SCT)
* Patients with previously untreated AML, MDS, or CMML-t who are considered inappropriate candidates for, or refused, standard induction chemotherapy due to older age or concurrent medical conditions are eligible
* No known CNS disease
* Performance status - ECOG 0-2
* See Disease Characteristics
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 5 times ULN
* Creatinine < 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to XK469R
* No other uncontrolled illness
* HIV-positive patients allowed provided CD4 counts are normal with no AIDS-defining disease
* No prior allogeneic SCT
* No concurrent prophylactic hematopoietic colony-stimulating factors
* More than 7 days since prior cytotoxic chemotherapy (except hydroxyurea)
* More than 7 days since prior radiotherapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anti-leukemia agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-10; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
MTD as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 21 days
Dose-limiting toxicity (DLT) defined as a clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications using CTCAE version 3.0 | 21 days

SECONDARY OUTCOMES:
Pharmacokinetic profile of XK496R | At baseline, at 15 and 30 minutes, and at 1, 2, 4, 6, 8, and 24 hours (of days 1-2), and at days 3 and 5
Candidate genes for XK469R using PCR assay | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Francis Giles, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States